CLINICAL TRIAL: NCT03294096
Title: Clinical Validation of Nutritional Supplements Developed for Pancreaticobiliary Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2017-0625
Record Dates: First submitted 2017-09-18; First posted 2017-09-26 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Pancreaticobiliary Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Dietary Supplement: Routine care + Nutritional product
- control group (Active Comparator)
  Interventions: Other: Routine care

INTERVENTIONS:
Dietary Supplement: Routine care + Nutritional product — Routine post-op care + Nutritional supplement by specific product
  Arms: experimental group
Other: Routine care — Routine post-op care
  Arms: control group

SUMMARY:
Decreased bowel function and loss of appetite in patients who underwent pancreaticobiliary surgery contribute impaired nutritional status in postoperative period. It can also affect perioperative and oncologic outcomes negatively. Therefore it is important to improve nutritional status in postoperative period by supply tailor-made optimal diets. The investigators have developed customized postoperative diets and products for pancreaticobiliary cancer patients. The investigators expect that nutritional supplement for pancreaticobiliary patients will increase the food intake rate and contribute a improvement of perioperative outcomes and even oncologic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age more than 19)
* Pancreaticobiliary cancer patient who is scheduled pancreaticoduodenectomy or distal pancreatectomy
* Pancreatic cancer / Duodenal cancer / Distal bile duct cancer / Ampulla of Vater cancer

Exclusion Criteria:

* Patient who denied clinical trial
* Diabetes Mellitus(DM) patient with DM complication
* Hyperlipidemia patient with vascular co-morbidity
* Impaired renal function or renal failure (GFP<70%)
* Poor nutritional status (PG-SGA grade C)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

PRIMARY OUTCOMES:
Food Intake Rate(%) for postoperative diet | Pre-operation
  Diet Intake Rate(%)
Food Intake Rate(%) for postoperative diet | 1 day before discharging
  Diet Intake Rate(%)
Food Intake Rate(%) for postoperative diet | 1 week after discharging (first outpatient follow up)
  Diet Intake Rate(%)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Hepatobiliary and Pancreatic Surgery, Department of Surgery, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided